CLINICAL TRIAL: NCT05141266
Title: Healthy Opioid Prescription Engagement 2.0
Brief Title: Healthy Opioid Prescription Engagement
Acronym: HOPE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jerry Cochran (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Jerry Cochran, Associate Professor, Internal Medicine, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 141016
Record Dates: First submitted 2021-11-08; First posted 2021-12-02 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Opioid Misuse; Opioid-Related Disorders; Pharmacist-Patient Relations
Keywords: Community Pharmacies; Patient Navigation; Opioid intervention
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Intervention Medication Therapy Management (BI-MTM) (Experimental): Brief Intervention Medication Therapy Management (BI-MTM) is the overarching model made up of 4 evidence-based components: Medication Therapy Management (MTM); Screening, Brief Intervention, and Referral to Treatment (SBIRT); naloxone dispensing, and Patient Navigation (PN). Each component is sequentially delivered within the model and addresses a critical aspect of opioid medication misuse and risk. The pharmacy-based portion of BI-MTM (MTM+SBIRT+naloxone) will be delivered by a PharmD level pharmacist, and PN will be delivered by a bachelor's level interventionist.
  Interventions: Behavioral: Patient Navigation
- Standard of Care (Other): Standard of Care is the treatment as usual condition, which follows federal and Utah state pharmacy requirements for pharmacists where in patients filling prescriptions receive information and opt-in counseling. Specifically, SMC in Utah requires pharmacists to: (1) offer counseling, (2) document counseling has been offered, (3) offer a counseling process for patients not present, and (4) discuss generic substitution.The duration of SMC in the current study is a single 5-10 minute session delivered by a University of Utah pharmacist other than the study pharmacist that possesses a similar level of education and professional licensing.
  Interventions: Other: Standard Medication Counseling (SMC)

INTERVENTIONS:
Behavioral: Patient Navigation — PN involves 8 weekly telephonic sessions lasting 30-45 minutes (telephonic to support lower-costs/sustainability). In session 1, the navigator reviews with the participant a report of scores from the baseline assessment to understand the participant's current health needs/challenges; session 1 also involves development of therapeutic alliance/rapport and goal setting. Sessions 2-4 focus on goal setting and identifying barriers and problem resolutions. The navigator elicits motivation and discusses this in context of readiness to change heath behavior and self-management skills. Sessions 2-4 also involve navigators supporting/assisting patients to fill out paperwork and enroll in needed social services and/or mental/behavioral/physical healthcare, including but not limited to primary care. Sessions 5-7 focus on encouraging and reinforcing treatment adherence, review-ing and identifying other care needs, and offering linkages to service providers as applicable
  Arms: Brief Intervention Medication Therapy Management (BI-MTM)
Other: Standard Medication Counseling (SMC) — SMC participants receive a single medication information/counseling session delivered by a University of Utah pharmacist to: (1) offer counseling, (2) document counseling was offered, (3) offer a counseling process for patients not present (not applicable to this study given all patients must screen in person), and (4) discuss generic substitution.
  Arms: Standard of Care

SUMMARY:
This study is a randomized controlled trial across 14 community pharmacies to test the efficacy of the Brief Intervention-Medication Therapy Management intervention (BI-MTM). The establishment of the BI-MTM model will result in a major impact for addressing the opioid epidemic, preventing opioid use disorder and overdose, and safeguarding patient health in a novel community-based service setting.

DETAILED DESCRIPTION:
This study examines a community pharmacy-based intervention to reduce opioid medication misuse. Despite a recent national decline in opioid prescribing, 10.3 million Americans in 2018 reported misusing a prescribed opioid, and within this population, >36% of those who misused obtained the opioid medication by filling a prescription. The point of medication dispensing, namely, the community pharmacy, is an untapped resource to address prescription opioid misuse-especially when considering the >60,000 pharmacies employing >170,000 pharmacists in the US. This study aims to conduct a fully-powered RCT of the BI-MTM intervention in community pharmacy settings that will accomplish 3 Specific Aims. The first Aim will demonstrate the pharmacist-led BI-MTM intervention is superior to standard medication counseling (SMC) for mitigating opioid medication misuse. This will be accomplished by conducting a powered single-blinded randomized trial to test the efficacy of BI-MTM (n=175) vs. SMC (n=175). Participants will be screened/recruited for eligibility at point of dispensing in 14 community pharmacies in Utah, a high opioid prescribing and opioid-adverse event state. Participants will be assessed at baseline, 2, and 6 months for opioid medication misuse. Participant-level state prescription drug monitoring data will also be linked with patient outcomes to assess objective changes in medication misuse behaviors (e.g., early refills and doctor/pharmacy shopping). The second Aim will identify the pathway by which BI-MTM results in improvements for depression, pain, and subsequently opioid misuse. To accomplish this, a path analysis will assess relationships of BI-MTM: (1) on depression, pain, and misuse, (2) depression on misuse, and (3) pain on misuse. The final Aim will explore latent transitions of baseline to post-intervention misuse classes by intervention group. This will be accomplished by using mixture modeling, specifically multi-group latent transition analysis. The observed misuse indicators will be used to estimate latent class transitions across time, grouping by treatment condition and adjusting for baseline covariates. Completing SA1- 3 advance the understanding of BI-MTM efficacy and set the stage for a national multisite trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* English speaking
* Not receiving cancer treatment
* Who have a positive opioid misuse screen on the POMI will be eligible to learn about this study

Exclusion Criteria:

* Are pregnant (given potential pre/post-natal opioid use complications among pregnant women/offspring
* Can-not provide collateral contact information for ≥2 contact persons (to ensure consistent contact/follow up)
* Do not have a reliable land line or mobile phone to be contacted by study staff
* Are filling only buprenorphine (given some formulations are not indicated for pain)
* Plan to leave the area for an extended period of time in the next 6 months
* Have had a psychotic and/or manic episode in the last 30 days (before consent, patients will be asked to screen for psychosis
* Do not provide permission to access their state prescription drug monitoring data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in opioid medication misuse. | 6 months
  This outcome will be assessed using the Prescription Opioid Misuse Index (POMI).

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Cochran, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cochran G, Shen J, Cox N, Field C, Carlston K, Sengpraseut B, White A, Okifuji A, Jackman C, Haaland B, Ragsdale R, Gordon AJ, Tarter R. Addressing opioid medication misuse at point of service in community pharmacy: A study protocol for an interdisciplinary behavioral health trial. Contemp Clin Trials. 2022 May;116:106759. doi: 10.1016/j.cct.2022.106759. Epub 2022 Apr 11. PMID 35417771